CLINICAL TRIAL: NCT06261437
Title: Effect of Ration Formulations on Warfighter Energy Balance and Physical Performance During a Field Training Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: M-11053; MO230060 (Other Grant/Funding Number: Military Operational Medicine Research Program (MOMRP))
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Close Combat Assault Ration (Experimental): The CCAR will be consumed as the sole nutrition source during a 7-day physically demanding military training exercise
  Interventions: Other: CCAR
- First Strike Ration (Active Comparator): The FSR will be consumed as the sole nutrition source during a 7-day physically demanding military training exercise
  Interventions: Other: FSR

INTERVENTIONS:
Other: CCAR — The CCAR will be consumed as the sole source of nutrition during a 7-day military training exercise.
  Arms: Close Combat Assault Ration
Other: FSR — The FSR will be consumed as the sole source of nutrition during a 7-day military training exercise.
  Arms: First Strike Ration

SUMMARY:
The goal of this randomized clinical trial is to determine the effects of consuming the Close Combat Assault Ration (CCAR) compared to the First Strike Ration (FSR) during a 7-day strenuous military training on energy intake and energy balance in healthy, Active Duty Warfighters.

The main questions it aims to answer are:

* Will consuming the CCAR result in lower energy intake or energy balance compared to consumption of the FSR?
* Will consuming the CCAR result in lower lower body strength or anaerobic power compared to consuming the FSR?
* Will those consuming the CCAR report lower ration acceptability or greater gastrointestinal side effects compared to those consuming the FSR?

Participants will be asked to consume either the CCAR or FSR as the sole nutrition source during a 7-day field training exercise (FTX). The vertical jump test, running-based anaerobic sprint test, and lower-body strength pull will be conducted pre and post the 7-day FTX to assess physical performance. Energy expenditure and intake will be measured by the doubly-labelled water method and dietary logs, respectively. Surveys will be completed to assess ration acceptability and gastrointestinal symptoms.

Researchers will compare the CCAR and FSR groups to see if their consumption impacted energy intake, energy balance, physical performance, ration acceptance, or gastrointestinal side effects.

DETAILED DESCRIPTION:
Army modernization priorities have identified the need to build the "capability to sustain multiple Brigade Combat Teams for up to seven days without periodic resupply to support semi-independent operations". To address this challenge and meet modernization requirements, ration developers from the Combat Feeding Division (CFD), Soldier Sustainment Directorate, Combat Capabilities Development Command - Soldier Center (DEVCOM-SC) developed the next generation ration, the Close Combat Assault Ration (CCAR). The CCAR is produced using novel food processing techniques that reduce weight and volume by removing air and water and increase the energy density by increasing the relative fat content. The result is a lightweight, low volume, energy-dense, shelf-stable, daily combat assault ration that provides Warfighters with meals that can be consumed while on the move, requiring no heating and little to no field preparation.

The ration will provide approximately 2800 kcals/day (47% carbohydrate, 12% protein, 41% fat) and includes a greater distribution of energy from fat to enable a smaller logistic footprint than the First Strike Ration (FSR, 2800 kcals/d; 58% carbohydrate, 12% protein, 30% fat).

This proposed project will evaluate the CCAR relative to the current recommended materiel solution (i.e., the FSR) in a field setting that approximates the operational conditions under which the ration will be consumed. Specifically, the proposed effort will compare energy intake, energy balance, physical performance, appetite, ration acceptability, and gastrointestinal responses in military personnel randomized to consume the CCAR or FSR in a multi-day training environment.

Participants will be randomized to consume the CCAR or FSR during a 7-day field training exercise. Physical performance will be assessed PRE and POST by the Running-Based Anaerobic Sprint Test, lower-body strength pull, and vertical jump. A subset of participants will consume doubly-labeled water and provide urine samples throughout the study period to measure energy expenditure. Appetite, ration acceptability, and gastrointestinal symptoms will be assessed by daily surveys. Energy intake will be measured by review of uneaten ration products and daily logs.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty male or female military personnel who are actively participating in the 7-day strenuous military training exercise.
* Willing to consume only foods/beverages provided by study staff during the training exercise, except for coffee and water.

Exclusion Criteria:

* Any injury or health condition limiting full participation in the 7-day Field Training Exercise.
* Any food allergy, lactose intolerance, or vegetarian practices.
* Not willing to participate in all study procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Energy intake | From study day 1 through 7
  Energy intake will be measured with daily food records and a review of food waste.
Energy expenditure | From baseline to study day 7
  Energy expenditure will be measured using the doubly-labeled water method.
Energy balance | From baseline to study day 7.
  Energy balance will measure the difference between energy intake and expenditure.

SECONDARY OUTCOMES:
Physical performance (vertical jump) | At baseline (PRE) and POST the 7-day FTX (i.e., study day 8)
  The maximum height of the vertical jump will be measured in cm.
Physical performance (peak power) | At baseline (PRE) and POST the 7-day FTX (i.e., study day 8)
  Peak power will be calculated from the vertical jump measure using the following equation:
  Peak Power (Watts) = [60.7 x jump height (cm)] + [45.3 x body mass (kg)] - 2055
Physical performance (Anaerobic capacity) | At baseline (PRE) and POST the 7-day FTX (i.e., study day 8)
  Anaerobic capacity will be measured by the time to complete the Running-Based Anaerobic Sprint Test.
Physical performance (lower-body strength) | At baseline (PRE) and POST the 7-day FTX (i.e., study day 8)
  Lower-body isometric strength will be measured using a Takei Back and Leg Dynamometer. The maximum strength (kg) during three trials will be used for analysis.
Food acceptance scale | From study day 1 through 7
  Food acceptance will be measured using a version of the Food Action Rating Scale. The Food Action Rating Scale is a Likert scale that measures food acceptance on a scale of 1-9. The scale ranges from dislike extremely (1) to like extremely (9).
Gastrointestinal Quality of Life Index | From baseline to study day 8
  Gastrointestinal quality of life will be measured using a modified version of the Gastrointestinal Quality of Life Index (GIQLI). Ratings of abdominal bloating, pain, nausea, and gastrointestinal discomfort will be assessed using a 100mm visual analog scale with values corresponding a range of symptoms (0; no symptoms to 100; extremely severe). The sum of the scores will represent GIQLI.
Hunger and Satiety Visual Analog Scales | From baseline to study day 8
  Ratings of subjective appetite sensations will be measured using 100 mm visual analog scales (VAS). Subjective ratings of hunger, fullness, desire to eat, and capacity to eat will be annotated on a 100mm line ranging from none (e.g., 0; Not at all hungry) to extremely (e.g., 100; extremely full).

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Dawson, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margolis LM, Rood J, Champagne C, Young AJ, Castellani JW. Energy balance and body composition during US Army special forces training. Appl Physiol Nutr Metab. 2013 Apr;38(4):396-400. doi: 10.1139/apnm-2012-0323. Epub 2013 Apr 3. PMID 23713532
- [Background] Hoyt RW, Jones TE, Baker-Fulco CJ, Schoeller DA, Schoene RB, Schwartz RS, Askew EW, Cymerman A. Doubly labeled water measurement of human energy expenditure during exercise at high altitude. Am J Physiol. 1994 Mar;266(3 Pt 2):R966-71. doi: 10.1152/ajpregu.1994.266.3.R966. PMID 8160893
- [Background] Karl JP, Hatch-McChesney A, Allen JT, Fagnant HS, Radcliffe PN, Finlayson G, Gwin JA, Margolis LM, Hennigar SR, McClung JP, Pasiakos SM. Effects of energy balance on appetite and physiological mediators of appetite during strenuous physical activity: secondary analysis of a randomised crossover trial. Br J Nutr. 2021 Nov 28;126(10):1571-1584. doi: 10.1017/S0007114521000131. Epub 2021 Jan 14. PMID 33441218

DOCUMENTS (1):
  • Informed Consent Form (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT06261437/ICF_000.pdf